CLINICAL TRIAL: NCT00776828
Title: Influence of CILostazol-based Triple Anti-platelet Therapy ON Ischemic Complication After Drug-eluting stenT Implantation
Brief Title: The Efficacy of CILostazol ON Ischemic Complications After DES Implantation
Acronym: CILON-T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyo-Soo Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CILON-T
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: cilostazol; clopidogrel; statin; drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAT (Active Comparator): triple antiplatelet therapy : aspirin, clopidogrel and cilostazol
  Interventions: Drug: cilostazol
- DAT (Placebo Comparator): dual antiplatelet therapy : aspirin, clopidogrel
  Interventions: Drug: cilostazol

INTERVENTIONS:
Drug: cilostazol — Pletaal (Otsuka Pharm.) 100mg bid for six months
  Other Names: Pletaal (Otsuka pharmaceutical)

SUMMARY:
Objectives :

* To evaluate the influence of concomitant use of cilostazol with aspirin and clopidogrel on the composite cardiovascular adverse outcomes (cardiac death, myocardial infarction, nonhemorrhagic stroke, target lesion revascularization) after drug-eluting stent implantation

Study Design : Prospective, open label, two arm, randomized multicenter trial to test the superiority of cilostazol group compared with the control group. Patients will be randomized according to the use of cilostazol

Patient Enrollment: 960 patients enrolled at 5 centers in Korea

Patient Follow-up : Clinical follow-up will occur at 1, 3 and 6 months. Angiographic follow-up will be recommended to all patient at 6 months after index procedure.

Primary Endpoint

* Composite of adverse cardiovascular/cerebrovascular outcomes (cardiac death, myocardial infarction, nonhemorrhagic stroke, target lesion revascularization) within 6 months

Secondary Endpoint

* All cause of death, stent thrombosis, and each component of primary endpoint at six months
* PRU level measured at discharge after the index procedure and after six months

Safety Endpoint

* Bleeding complications according to TIMI criteria
* The incidence of drug discontinuation
* Heart rate

DETAILED DESCRIPTION:
Stratified randomization by statin type (rosuvastatin or atorvastatin) and the center was performed

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at leat 18 years of age
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of cilostazol and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have significant coronary artery stenosis (>50% by visual estimate)
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or reversible changes in the electrocardiogram (ECG) consistent with ischemia. In subjects with coronary artery stenosis>75%, evidence of myocardial ischemia does not have to be documented.
* Coronary lesions must be amenable for percutaneous coronary revascularization with drug eluting stents.

Exclusion Criteria:

* Subject who undergoes primary percutaneous coronary intervention due to acute ST elevation myocardial infarction
* Subject who has contraindication or allergy to anti-platelet agents (aspirin, clopidogrel or cilostazol)
* Subject who has thrombocytopenia (<120,000/uL)
* Subject who has liver cirrhosis (Child class B or C)
* Subject who is on the anticoagulation therapy
* Subject who has severe congestive heart failure (left ventricular ejection fraction <30%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Composite of adverse cardiovascular outcomes | six months
  composite of cardiac death, myocardial infarction, ischemic stroke and target lesion revascularization

SECONDARY OUTCOMES:
all cause of death | six months
stent thrombosis | six months
each component of primary endpoint | six months
PRU level | at discharge after the index procedure
PRU level | six months after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD,PhD, Principal Investigator — Seoul National University Hospital; In-Ho Chae, MD, PhD, Study Chair — Seoul National University Bundang Hospital; Jang-Ho Bae, MD, PhD, Study Chair — Gonyang University Hospital; Myung-Chan Cho, MD, PhD, Study Chair — Chungbuk National University Hospital; Seung-Woon Rha, MD, PhD, Study Chair — Korea University Guro Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Suh JW, Lee SP, Park KW, Lee HY, Kang HJ, Koo BK, Cho YS, Youn TJ, Chae IH, Choi DJ, Rha SW, Bae JH, Kwon TG, Bae JW, Cho MC, Kim HS. Multicenter randomized trial evaluating the efficacy of cilostazol on ischemic vascular complications after drug-eluting stent implantation for coronary heart disease: results of the CILON-T (influence of CILostazol-based triple antiplatelet therapy ON ischemic complication after drug-eluting stenT implantation) trial. J Am Coll Cardiol. 2011 Jan 18;57(3):280-9. doi: 10.1016/j.jacc.2010.08.631. PMID 21232664
- [Derived] Lee SP, Suh JW, Park KW, Lee HY, Kang HJ, Koo BK, Chae IH, Choi DJ, Rha SW, Bae JW, Cho MC, Kwon TG, Bae JH, Kim HS; CILON-T investigators. Study design and rationale of 'Influence of Cilostazol-based triple anti-platelet therapy on ischemic complication after drug-eluting stent implantation (CILON-T)' study: A multicenter randomized trial evaluating the efficacy of Cilostazol on ischemic vascular complications after drug-eluting stent implantation for coronary heart disease. Trials. 2010 Aug 24;11:87. doi: 10.1186/1745-6215-11-87. PMID 20735821